CLINICAL TRIAL: NCT06043206
Title: Bariatric Surgery in Patients With Schizophrenia
Acronym: SCHIZOBAR
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Hospital del Mar (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government); Parc Taulí Hospital Universitari (Other); University Hospital A Coruña (Other); Hospital General Universitario Gregorio Marañon (Other); University of Navarrra Hospital (Clinica Universitaria) (Other); Hospital Clinic of Barcelona (Other); León University Assistance Complex, Leon, Spain (Unknown); Valle del Nalón Hospital, Asturias, Spain (Unknown); Complejo Hospitalario Universitario de Vigo (Other); Hospital Arnau de Vilanova (Other); Hospital San Carlos, Madrid (Other); Hospital Universitari de Bellvitge (Other); Hospitales Universitarios Virgen del Rocío (Other); Hospital Regional de Malaga (Other); Germans Trias i Pujol Hospital (Other); Hospital Universitario Virgen Macarena (Other); Hospital Mutua de Terrassa (Other); Hospital Son Llatzer (Other); University Hospital of Girona Dr. Josep Trueta (Network); University Hospital of the Canary Islands, Tenerife, Spain (Unknown); Hospital Virgen de la Luz (Other); Hospital Universitario Virgen de la Victoria (Other); Viladecans Hospital, Barcelona, Spain (Unknown); Hospital Universitario Doctor Peset (Other); Hospital Universitari Sant Joan de Reus (Other); General Hospital, Vic, Spain (Unknown)
Responsible Party: Sponsor
Other Study IDs: IIBSP-BAR-2022-30
Record Dates: First submitted 2023-09-03; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Obesity; Schizophrenia
Keywords: Bariatric Surgery; Hospital care; Observational study; weight loss; evolution
MeSH Terms: conditions — Obesity; Schizophrenia; Weight Loss | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases Obesity and schizophrenia: Patients with schizophrenia and obesity undergoing bariatric surgery
  Interventions: Procedure: Bariatric Surgery
- Controls: Patients without psychiatric pathology matched by age, sex, BMI and type of surgery and in a 4:1 ratio to cases.
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Procedure: Bariatric Surgery — Bariatric Surgery

SUMMARY:
It is known that schizophrenia is associated with obesity in a significant number of patients and it implies a poor prognostic factor, with weight loss being important in this population. However, data about the prognosis of weight loss surgery in subjects with schizophrenia is scant.

Hypothesis: Bariatric surgery in subjects with schizophrenia leads to an improvement in weight and cardiometabolic comorbidities similar to that of subjects without schizophrenia Main goal: To study the evolution after bariatric surgery in patients with obesity and schizophrenia Design: Multicenter retrospective case control study. Disease under study: Schizophrenia and Obesity Methodology: Retrospective observational study Study population and total number of subjects Cases: Patients with schizophrenia and obesity undergoing bariatric surgery. (number: all cases collected within the GOSEEN group).

Controls: Patients without psychiatric pathology matched by age, sex, body mass index and type of surgery and in a 4:1 ratio to cases.

Calendar. Expected duration of the study. 12 months ethical considerations Informed consent will be obtained from patients who are currently being followed up at the reference centers.

DETAILED DESCRIPTION:
THEORETICAL FRAMEWORK. PROBLEM STATEMENT:

Background Obesity affects approximately 45-55% of patients with schizophrenia (1). Weight gain in these patients may be due to different factors such as the use of antipsychotic drugs with an unfavorable metabolic profile, the coexistence of sleep disorders or negative cognitive symptoms that often translate into a more sedentary lifestyle and alterations in eating behavior, among others (2). The coexistence of obesity and its comorbidities in this group of patients significantly worsens both their physical and mental health (3). In fact, cardiovascular disease is one of the main causes of mortality in patients with schizophrenia (4).

Lifestyle interventions, while they may be effective in people with schizophrenia (5), often fall short of achieving weight goals. At present, obesity surgery represents the most effective treatment in terms of weight loss and resolution of comorbidities, being indicated in cases of patients with a body mass index (BMI) > 35 kg/m2 with comorbidities or BMI > 40 Kg/m2 with/without comorbidities. However, the access of patients with schizophrenia to bariatric surgery techniques is usually limited by different factors such as fear of a possible worsening of the underlying disease, or a lower weight loss in this population, among others. In addition, clinical practice guidelines recommend that all patients with psychiatric pathologies be evaluated in a regulated manner prior to surgery (6), although the content of this evaluation and the criteria for declining or accepting surgery are not clear. Although the course of schizophrenia is variable and its symptoms may be stable without being a clear contraindication for bariatric surgery, in actual practice, a considerable number of professionals contraindicate bariatric surgery in the presence of a psychotic disorder (7).

For these reasons, data on the efficacy of bariatric surgery in patients with schizophrenia are scarce and limited to very small case series with short-term follow-up (2,8,9). Our objective is therefore to carry out a multicenter retrospective study that allows us to study the long-term evolution after bariatric surgery in a large series of patients, focusing not only on weight evolution but also on the long-term evolution of psychiatric pathology.

Justification It is necessary to have information about the prognosis of subjects with severe obesity and schizophrenia who undergo bariatric surgery. This knowledge will make it possible to establish clear guidelines for action in these cases.

Research questions What is the long-term outcome after bariatric surgery in subjects with schizophrenia? Hypothesis Bariatric surgery in subjects with schizophrenia leads to an improvement in weight and cardiometabolic comorbidities similar to that of subjects without schizophrenia

GOALS:

Main goal:

To study the short (first year after bariatric surgery) and long-term (up to 5 years of follow-up after bariatric surgery) evolution in terms of weight loss of patients with obesity and schizophrenia who underwent bariatric surgery in Spain and compare it with the evolution of patients without psychiatric disorder.

Secondary objectives:

* Determine the casuistry of patients, with special interest in the characteristics of the underlying psychiatric pathology (years of evolution, clinical stability criteria, pharmacological treatment...).
* To Analyze the evolution of obesity comorbidities.
* To Analyze the evolution of psychiatric pathology after bariatric surgery: (decompensation, drug treatment...)
* To analyze the frequency of early (<30 days post-surgery) or late (>30 days post-surgery) post-surgical complications.

METHODS:

Study design Retrospective case-control study.

Expected sample size All cases detected in Spanish territory The minimum number of cases expected will be 10 patients based on the low casuistry of the problem. The number of patients in the control group will be x4 that in the study group.

Methodology. Information sources The study population will be identified in each center in the usual specialty consultations or by searching the databases of each center. Review of medical records in search of the specified variables (retrospective observational study).

Data Management and Analysis The coordinating researcher (Dra Inka Miñambres Donaire) will be responsible for the creation of the database and its exploitation. The database will be created in Excell format and the SPSS program will be used for statistical analysis. The statistics will be mainly descriptive. For cases in which it is decided to compare groups, normality tests will be used to establish the behavior of the variables and parametric/non-parametric tests will be used as appropriate.

Data collection The researcher will guarantee the accuracy and integrity of the data, as well as all the reports that are required. The data included in the Data Collection Notebook (CRD), which are derived from source documents, will be consistent with those documents or otherwise the discrepancies will be justified.

The researcher will keep the study documents until at least 5 years after completion.

At the request of the monitor, auditor, ethics committee or health authority, the researcher will have available all the files related to the study, allowing direct access to the data or source documents for monitoring, auditing, review by the ethics committee, as well as the inspection of the trial by the competent authorities.

Limitations of the design, the source of information and the methods of analysis

The main limitation of the study is its retrospective nature. However, the study design is adequate given the low frequency of the pathology.

Data confidentiality Regarding the confidentiality of the study data, the provisions of Organic Law 3/2018, of December 5, on the Protection of Personal Data and Guarantee of Digital Rights and the General Regulation (EU) on Data Protection will be followed. 2016/679.

Interference with physician's prescribing habits As it is a retrospective study, there will be no interference with the prescribing habits of the doctor.

ELIGIBILITY:
Cases:

Inclusion) Both criteria must be met:

1. Patients with severe obesity undergoing bariatric surgery and with follow-up in Spanish territory.
2. Patient with schizophrenia or schizoaffective disorder.

Exclusion) Subjects who do not meet any of the two inclusion criteria

Controls: in a 4:1 ratio with cases

Inclusion) Both criteria must be met:

1. Patients with severe obesity undergoing bariatric surgery and with follow-up in Spanish territory.
2. Absence of psychiatric pathology
3. Paired with the cases by age, sex, BMI before surgery and type of surgery.

Exclusion) Subjects who do not meet any of the two inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: subjects undergoing bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Weight loss | 12 months and 5 years after the surgery
  short (first year after bariatric surgery) and long-term (up to 5 years of follow-up after bariatric surgery) evolution in terms of weight loss of patients with obesity and schizophrenia who underwent bariatric surgery

SECONDARY OUTCOMES:
Clincial Caracteristics description | inclusion, day 1
  casuistry of patients, with special interest in the characteristics of the underlying psychiatric pathology (years of evolution, clinical stability criteria, pharmacological treatment...)
Comorbidity progression | 12 months and 5 years after the surgery
  Analyze the evolution of obesity comorbidities: presence of type 2 diabetes, hypertension, OSAS and dyslipidemia. Remission of co morbidities was defined as cessation of medication for hypertension or hyperlipidemia with normal blood pressure and lipid levels, cessation for continuous positive pressure ventilation for sleep apnea, and normalization of HbA1C (<6.5) with no medications for diabetes.
Psychiatric pathology progression | 30 days post surgery and 5 years after the surgery
  Analyze the evolution of psychiatric treatment: Psychiatric medication burden will be calculated by generating a continuous variable using a previous validated formula (Central Nervous System Medication Burden and Serious Falls in Older Nursing Home Residents Joseph T. Hanlon, J Am Geriatr Soc. 2017 June ; 65(6): 1183-1189. doi:10.1111/jgs.14759).
post-surgical complications | up to 30 days post-surgery) or late post-surgical complications (through study completion, up to five years post-surgery)
  To analyze the frequency of early or late post-surgical complications

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
individual participant data can not be available due to the data protection law restrictions, however, anonymized data could be shared on demand

DOCUMENTS (2):
  • Study Protocol (2022-02-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT06043206/Prot_000.pdf
  • Informed Consent Form (2022-02-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT06043206/ICF_001.pdf